CLINICAL TRIAL: NCT05228808
Title: Prognostic Value of Immunohistochemical Expression of PD-L1 in Pancreatic Ductal Adenocarcinoma
Brief Title: Immunohistochemical Expression of PD-L1 in Pancreatic Ductal Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nagwa Abd El-Sadek Ahmed, Lecturer at Pathology Department, Faculty of Medicine, Sohag University, Sohag University
Other Study IDs: Soh-Med-22-01-30
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic ductal adenocarcinoma; PD-L1; Prognostic value

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic carcinoma is ranked the 11th most common cancer worldwide. It is a highly lethal malignant tumor. In Egypt, the disease has traditionally been considered rare, but population in the East Nile Delta region exhibits an unusually high rate of young-onset pancreatic carcinoma. Pancreatic ductal adenocarcinoma is by far the most common histologic subtype of pancreatic malignancy. Programmed death ligand-1 (PD-L1) is a type I trans-membrane glycoprotein. It has an important prognostic and predictive value in various neoplasms. To date, few studies have addressed the potential prognostic role of PD-L1 in pancreatic carcinoma, so knowledge about its prognostic value needs further elucidation.

DETAILED DESCRIPTION:
Pancreatic carcinoma is ranked the 11th most common cancer worldwide. It is a highly lethal malignant tumor with 5-year survival rate as low as 9%. It is the seventh leading cause of cancer-related deaths both in men and women worldwide. In Egypt, the disease has traditionally been considered rare, but population in the East Nile Delta region exhibits an unusually high rate of young-onset pancreatic carcinoma.

Pancreatic ductal adenocarcinoma is by far the most common histologic subtype of pancreatic malignancy, accounting for about 90% of all pancreatic malignant neoplasms. Hence, the terms "pancreatic cancer" and "pancreatic ductal adenocarcinoma" are often used synonymously. Most pancreatic adenocarcinomas occur in the head of pancreas; about 60-70%. Tobacco smoking, diabetes mellitus, obesity, alcohol consumption, family history, certain genetic polymorphisms and chronic pancreatitis have been considered as risk factors for pancreatic adenocarcinoma.

Pancreatic adenocarcinoma typically has a very poor prognosis. Although therapeutic strategies have been developed in recent years, the prognosis isn't significantly improved. To date, a group of prognostic factors are identified for clinical management of pancreatic adenocarcinoma. However, these markers are lack of accuracy to predict the outcome and aren't widely adopted. Therefore, it is still important to find out novel prognostic and predictive biomarkers to explore promising fields of research in terms of treatment selection and tailored therapy in pancreatic carcinoma.

Immunotherapy is a rapidly growing field and represents a paradigm shift in the treatment of malignant tumors; it has made clinically significant breakthroughs in the last decade. Targeting immune checkpoints has had immense clinical success resulting in sustained treatment response for a subset of patients with certain malignancies. Currently, many clinical trials seek to assess the efficacy of immunotherapeutic strategies in pancreatic adenocarcinoma.

Programmed death ligand-1 (PD-L1) is a type I trans-membrane glycoprotein. It acts as a ligand for Programmed death-1 (PD1) and has an important prognostic and predictive value in various types of neoplasms. It is overexpressed in several neoplasms such as bronchogenic carcinoma, hepatocellular carcinoma and breast cancer. PD1 and PD-L1 are immune checkpoints and members of cytotoxic T lymphocyte antigen-4 family. They are responsible for immunosuppression and decreased antitumor cytokines. They are expressed by tumor cells to escape immune surveillance. Moreover, PD1/PD-L1 pathway activates the intercellular signals that inhibit apoptosis and enhance survival of tumor cells. PD1 and PD-L1 are targeted in many clinical trials; blockade of the immune checkpoints activated by the PD-1/PD-L1 pathway has demonstrated impressive benefits in various neoplasms such as melanoma and non-small cell lung cancer.

Blockade of PD-L1 is a prevalent strategy of cancer immunotherapy; the use of checkpoint inhibitors to target the PD1/PDL1 pathway results in breakthrough in the immunotherapy field. A number of studies investigated the association of PD-L1 and prognosis of pancreatic carcinoma, with controversial results presented [8]. To date, few studies have addressed the potential prognostic role of PD-L1 in pancreatic carcinoma, so knowledge about its prognostic value needs further elucidation.

The aim of this study is to evaluate the expression of PD-L1 in pancreatic ductal adenocarcinoma and to correlate its expression to different studied histopathological parameters to evaluate its prognostic value.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic ductal adenocarcinoma who underwent surgery.

Exclusion Criteria:

* Patients received pre-operative chemotherapy or radiotherapy.
* Patients with insufficient clinical data.
* Specimens with extensive necrosis
* Tiny specimens which are insufficient for accurate diagnosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fifty specimens of pancreatic adenocarcinoma obtained from patients who underwent surgery, according to local Ethical Committee regulations, to be examined in the Pathology Laboratory of Sohag Faculty of Medicine. From January 2022 till completing the sample size.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the expression of PD-L1 in pancreatic ductal adenocarcinoma | 1 month
  Immunohistochemical study
correlate PD-L1 expression to different studied histopathological parameters to evaluate its prognostic value. | 1 month
  Statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Ahmed, Lecturer, Principal Investigator — Sohag University
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt